CLINICAL TRIAL: NCT02306980
Title: Oral Administration of Colostrum to Premature Babies: Impact on the Oral Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 531791
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Changes in the Oral Microbiota

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colostrum (Experimental): Colostrum administration
  Interventions: Other: Colostrum
- Control (No Intervention): Routine care

INTERVENTIONS:
Other: Colostrum — Mother's own colostrum (0.2 ml) will be administered into the mouth of the infant every 2 hours for 48 hours.
  Arms: Colostrum

SUMMARY:
Oropharyngeal administration of mother's colostrum to premature infants has been proposed as a stimulus to the oropharyngeal lymphatic tissues to decrease the incidence of pneumonia and sepsis, particularly in intubated babies. We propose to study the impact of this intervention on the composition of the oral microbiota.

ELIGIBILITY:
Inclusion Criteria:

* premature infant with birth weight < 1500
* intubated in the first 48 hours of life
* available maternal colostrum

Exclusion Criteria:

* lethal condition

Ages: 12 Hours to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2013-10; Primary Completion 2015-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Oral microbiota | Difference between enrollment, 48 hours and 96 hours
  Changes in the composition of the community of microbes inhabiting the oral-cavity after administration of oropharyngeal maternal colostrum.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Underwood, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Children's Hospital, Sacramento, California, United States

REFERENCES:
- [Derived] Sohn K, Kalanetra KM, Mills DA, Underwood MA. Buccal administration of human colostrum: impact on the oral microbiota of premature infants. J Perinatol. 2016 Feb;36(2):106-11. doi: 10.1038/jp.2015.157. Epub 2015 Dec 10. PMID 26658119